CLINICAL TRIAL: NCT05529745
Title: Neurorehabilitation Impact on Neurocognitive Impairments in Cerebellar Lesions
Acronym: NRCEcog
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Klinik Bavaria (Other)
Responsible Party: Principal Investigator, Michael Adamaszek, Michael Adamaszek, head of Dept. Clinical and Cognitive Neurorehabilitation, Klinik Bavaria
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: EK-BR-158/20-1
Record Dates: First submitted 2022-08-26; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Cerebellum; Injury
Keywords: Cerebellum - cognitive functions - neurorehabilitation
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment in cerebellar lesioned patient (Experimental): Group of patients with a lesion of the cerebellum gaining a neurorehabilitation intervention
  Interventions: Other: Neurorehabilitation cerebellar cognitive disorder
- Treatment in supratentorial lesioned patient (Active Comparator): Group of patients with a lesion of the supratentorial area gaining a neurorehabilitation intervention
  Interventions: Other: Neurorehabilitation cerebellar cognitive disorder

INTERVENTIONS:
Other: Neurorehabilitation cerebellar cognitive disorder — Influence of neurorehabilitation treatment lines of physiotherapy and exercise therapy including scheduled occupational therapy to adapt and improve cognitive-affective disorders in cerebellar lesions.

SUMMARY:
Depending on their localization, cerebellar lesions cause various pronounced cognitive and/or affective dysfunctions, which are causally related to the involvement of cerebellar structures in neuronal networks for higher-order processing of cognitive and emotional items in the association areas of the cerebral cortex. For further investigation, event-related potential (ERP) analyses will be performed to record and visualize specific signals in the surface EEG, which should provide information about the course of treatment of neurorehabilitation with respect to a close correlation and thus predictive power to functional recovery that occurred as a result of cerebellar injury. With EEG parameters and clinical examination findings including neuropsychology, the functions for four thematically distributed domains (affective: prosody; cognitive: abstraction, linguistic and formal incongruence) will be recorded and evaluated over a four-week structured neurorehabilitation with an average therapy volume.

DETAILED DESCRIPTION:
Cerebellar damage causes various cognitive and affective dysfunctions to varying degrees depending on its location, with cognitive abnormalities seen primarily in the posterior lobes, whereas disorders of affect modulation are seen more frequently in lesions of the vermis. Causally, cerebellar structures are thought to be involved in neuronal networks distributed primarily within temporal, parietal, and frontal association cortices for higher-order processing of cognitive and emotional items. Based on the evidence to date, cerebellar areas appear to be involved at the level of congruent and incongruent associations with different temporal binding of the cerebral networks responsible for them. For further investigation, event-related potential (ERP) analyses will be performed to capture and represent temporal signal dynamics in surface EEG, which will be used to calculate predictive values for the quality and extent of neurorehabilitation applications for functional recovery and thus clinical outcome via neurophysiological markers. In addition to clinical scales and neuropsychological investigations, the processing of four thematically distributed (prosody, abstraction, linguistic and formal incongruence) trials at the beginning and after about four weeks of a structured neurorehabilitation with a therapy volume of at least 20 hours per week of physical and occupational therapy as well as computer-assisted exercises, in their temporal and topographical characteristics of neurophysiologically tangible functional disorders and their dynamics in the course of treatment will be investigated via the derivation of ERP.

ELIGIBILITY:
Inclusion Criteria:

* active group: patients with a cerebrovascular lesion within the cerebellum
* comparator group: patients with a cerebrovascular lesion supratentorial

Exclusion Criteria:

* any kind of history in neurological or psychiatric disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Changes of attentional and executive functioning in active group. | 26 weeks
  Beneficial changes in attentional and executive function performance in ischemic cerebellar injury after structured neurorehabilitation modules. Measurements will be succeed by the Cerebellar Cognitive Affective/ Schmahmann Syndrome Scale (German version) with a maximum of 120 of 120 points, i.e. an increase of the test performance with higher point values along the neurorehabilitation procedure is considered as an indication of clinical improvement.

SECONDARY OUTCOMES:
Extension of daily activities and life quality. | 52 weeks
  Growing action behavior (recorded by SF-36 scale) in everyday life, whereby an increase from low point values up to high point values (between a range of 0 points with very low quality of life as minimum, and up to 100 points as a maximum of quality of life) indicates a growing quality of life due to neurologic impromenet .

IPD SHARING:
Plan to Share IPD: No